CLINICAL TRIAL: NCT00946010
Title: Investigation of Hepatitis B and Hepatitis C in Taiwan
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 200801059R
Record Dates: First submitted 2008-04-01; First posted 2009-07-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Hepatitis B; Hepatitis C
Keywords: Hepatitis B; Hepatitis C; genotype; DNA level; RNA level; Taiwan
MeSH Terms: conditions — Hepatitis B; Hepatitis C | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 10ml blood was sampled and then serum was be retained.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Click here for more information about this study: Investigation of Hepatitis B and Hepatitis C in Taiwan
  Interventions: Biological: blood sampling and abdominal sonography

INTERVENTIONS:
Biological: blood sampling and abdominal sonography — 10cc blood sampling and abdominal sonography
  Other Names: 10cc blood sampling and abdominal sonography

SUMMARY:
The purpose of this study is to investigate the differences of genotypes of hepatitis B and hepatitis C in Taiwan.

DETAILED DESCRIPTION:
The purpose of this study is investigating the differences of genotypes and DNA level or RNA level of hepatitis B and hepatitis C in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Born before 1985/01/01
* HBV or HCV carriers

Exclusion Criteria:

* N/A

Min Age: 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People Born before 1985/01/01 who live in Taiwan are HBV or HCV pateints.
Sampling Method: Non-Probability Sample
Enrollment: 6228 (Actual)
Dates: Start 2008-04; Primary Completion 2010-08 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
genotype and DNA level or RNA level of HBV and HCV virus | once during Mar. 2008- Jan. 2011

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Chuan Sheu, M.D. P.H.D., Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan